CLINICAL TRIAL: NCT00949507
Title: Comparison of Two Regimens of Anesthesia for Children Undergoing MRI in General Anesthesia. Advantages, Disadvantages and Time Consumption Regarding the Two Regimens.
Brief Title: Comparison of Two Regimens of Anesthesia for Children Undergoing Magnetic Resonance Imaging (MRI) in General Anesthesia
Status: Completed | Type: Observational
Sponsor: Niels Anker Pedersen (Other)
Responsible Party: Sponsor-Investigator, Niels Anker Pedersen, MD, Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Other Study IDs: 2008-209; EudraCT 2008-002690-12; 2008-41-2609; 2612-3762; H-A-2008-060
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: General Anesthesia; Children; MRI; Sevoflurane; Propofol/Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- anaesthesia using propofol: the children are anaesthetized using intravenous anaesthesia with propofol and remifentanil; a binasal catheter is used for administration of oxygen during the anaesthesia
- anaesthesia using sevoflurane: the patients are anaesthetized using sevoflurane 1 MAC; a laryngeal mask is used

SUMMARY:
Comparison of two regimens (Sevorane/LMA ctr. Propofol/Remifentanil) for children undergoing MRI in general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* children aged 1 to 10 yrs.
* ASA 1-2

Exclusion Criteria:

* Allergy to soya (propofol)
* Allergy to Pentobarbital
* Allergy to Remifentanil
* Allergy to Sevoflurane
* Children undergoing blood tests or further examinations in conjunction with the MRI
* Children with unexplained fever
* Children which are evaluated not to be able to keep a open airway

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 120 children ASA 1-2 aged 1 to 10 yrs. scheduled for MRI in general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
postanaesthetic recovery and behavioral score | 0-24 hours hours postoperatively

SECONDARY OUTCOMES:
Time span of the recovery process | 0-3 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup University Hospital, Dept. of Anesthesia, Glostrup Municipality, Copenhagen, Denmark